CLINICAL TRIAL: NCT01577433
Title: Driveline Silicone Skin Interface (SSI) Registry
Brief Title: Driveline Silicone Skin Interface Registry
Acronym: SSI
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TC11282011
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Driveline Heart-assisted Device Related Infection
Keywords: HeartMate II; heart-assist device; left ventricular assist device; driveline infection; LVAD; HMII LVAS driveline; silicone portion; Thoratec Corporation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: Historical control HeartMate II BTT and DT data
- Prospective and Retrospectively identified SSI: Prospectively and Retrospectively identified HeartMate II patients where the full length of the velour coated portion of the driveline is tunneled under the skin

SUMMARY:
The purpose of this observational registry is to determine the freedom from driveline (DL) infection events in subjects implanted with a HeartMate II LVAD in whom only the silicone portion of the DL is externalized resulting in a silicone skin interface (SSI)

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed the INTERMACS informed consent form
* Subject has signed the SSI registry informed consent form
* Subject age ≥ 18 years
* Subject implanted with a HeartMate II LVAD
* Subject in whom the full length of the velour portion of the percutaneous lead is fully kept under the skin resulting in a silicone skin interface at the skin exit site
* In the prospective study cohort, Subject is planned to be supported with the HeartMate II LVAD for at least 12 months
* In the retrospective study cohort, at the time of enrollment, Subject has been supported with a HeartMate II for at least 10 months

Exclusion Criteria:

* In the retrospective study cohort, Subject is ongoing with long-term right heart mechanical circulatory support (RVAD)
* In the retrospective study cohort, Subject had a post-implant sternal re-entry (for bleeding, etc.) or delayed sternal closure
* In the retrospective study cohort, Subject is participating in any other clinical investigation related to driveline (DL) exit site that could confound the study results
* In the prospective study cohort, Subject is participating in any other clinical investigation related to driveline (DL) exit site that could confound the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are implanted/have been implanted with the commercially available HeartMate II LVAD for approved indications
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-05; Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Freedom from DL infection events at 12 months after LVAD implantation | 12 Months

SECONDARY OUTCOMES:
Percentage of subjects with infection events | Month 1, 3, 6, and every six months up to 60 months post-enrollment
DL infection events per patient year | Month 1, 3, 6, and every 6 months up to 60 months post-enrollment
DL tunneling methods or other factors that might reduce risks of DL related infection events | Month 1, 3, 6, and every 6 months up to 60 months post-enrollment

CONTACTS AND LOCATIONS:
Overall Officials: David Farrar, PhD, Study Director — Abbott Medical Devices
Locations (15):
- United States (15):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St.Vincent's Hospital and Health Services, Indianapolis, Indiana
  - University of Iowa Hospital, Iowa City, Iowa
  - Henry Ford Hospital, Detroit, Michigan
  - Abbott Northwestern, Minneapolis, Minnesota
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Baylor Medical Center, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Sacred Heart Medical Center, Spokane, Washington

REFERENCES:
- [Background] Akhter SA, Ewald GA, Walsh MN, et al. Preliminary driveline infection results from the multicenter silicone-skin-interface (SSI) registry. Abstracts from the ASAIO 59th Annual Conference, p. 61. http://journals.lww.com/asaiojournal/Documents/ASAIO%20Abstracts%202013.pdf